CLINICAL TRIAL: NCT06185400
Title: Disitamab Vedotin（RC48）Combined With EGFR or HER2 TKI for Locally Advanced or Metastatic NSCLC Patients With HER2 Alterations
Brief Title: RC48 Combined With EGFR or HER2 TKI for Locally Advanced or Metastatic NSCLC Patients With HER2 Alterations
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jie Wang, Head of Oncology Department, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RCVDODIIR010
Record Dates: First submitted 2023-11-28; First posted 2023-12-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Non Small Cell Lung Cancer; ERBB2 Mutation-Related Tumors; ERBB2 Gene Duplication; Disitamab Vedotin
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — disitamab vedotin; aumolertinib; pyrotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm1: Treatment Naive NSCLC (Experimental): RC48+third-generation EGFR TKIs in treatment-naive patients harboring EGFR mutation and HER2 alterations
  Interventions: Drug: Disitamab Vedotin; Drug: third-generation EGFR TKIs (Almonertinib/Furmonertinib/Osimertinib)
- Arm2: Locally Progressed (Experimental): This cohort includes ERBB2 altered patients after third-generation EGFR-TKIs treatment with locally or slowly progressed disease, who may continue to benefit from third-generation EGFR-TKIs treatment under investigators' evaluation.
  Interventions: Drug: Disitamab Vedotin; Drug: third-generation EGFR TKIs (Almonertinib/Furmonertinib/Osimertinib)
- Arm3: Extensively Progressed (Experimental): This cohort includes ERBB2 altered patients after third-generation EGFR-TKIs treatment with extensively progressed disease, who may be less likely to benefit from third-generation EGFR-TKIs treatment under investigators' evaluation.
  Interventions: Drug: Disitamab Vedotin; Drug: pyrotinib

INTERVENTIONS:
Drug: Disitamab Vedotin — RC48+third-generation EGFR TKIs (Almonertinib/Furmonertinib/Osimertinib) in treatment naive NSCLC
  Other Names: RC48
Drug: third-generation EGFR TKIs (Almonertinib/Furmonertinib/Osimertinib) — RC48+third-generation EGFR TKIs (Almonertinib/Furmonertinib/Osimertinib) after EGFR-TKIs progression
  Arms: Arm1: Treatment Naive NSCLC; Arm2: Locally Progressed
Drug: pyrotinib — RC48+pyrotinib after EGFR-TKIs progression
  Arms: Arm3: Extensively Progressed

SUMMARY:
Disitamab Vedotin（RC48）combined with EGFR or HER2 TKIs in locally advanced or metastatic NSCLC Patients with HER2 Alterations.

DETAILED DESCRIPTION:
This study will explore the treatment of locally advanced or metastatic non-small cell lung cancer with HER2 mutation, amplification, or HER2 protein overexpression, using Disitamab Vedotin（RC48）combined with EGFR or HER2 TKIs, in the aim of providing new treatment strategies for lung cancer patients with HER2 pathway activation.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 (inclusive) or above, regardless of gender.
2. Histologically or cytologically confirmed locally advanced or metastatic NSCLC, not suitable for radical surgery or radiotherapy (TNM 8th Edition).".
3. HER2 alterations include HER2 gene mutations, gene amplification and HER2 protein over-expression;
4. Number of treatment lines:

   * Arm1: patients who have not previously received systemic treatment for advanced diseases;
   * Arm2: Previously received first line of third-generation EGFR-TKIs treatment with local progression, oligometastasis, or slow progression, and evaluated by the researchers to continue to benefit from third-generation EGFR-TKIs treatment;
   * Arm3: Previously received first line of third-generation EGFR-TKIs treatment with extensively progression, and evaluated by the researchers not likely to continue to benefit from third-generation EGFR-TKIs treatment;
5. There is at least one measurable lesion that meets the definition of the RECIST 1.1 standard at baseline.
6. ECOG fitness status score: 0 or 1 point.

Exclusion Criteria:

1. Central nervous system metastasis or meningeal metastasis with clinical symptoms.
2. Known hypersensitivity or intolerance to any component of the study protocol drug or its excipients.
3. Have a history of severe cardiovascular disease.
4. Have a history of interstitial lung disease or drug-induced interstitial lung disease requiring steroids treatment; radiation pneumonia.
5. Have a history of neurological disorders or mental illnesses, including epilepsy or dementia.
6. Pregnant or lactating women.
7. The researcher believes that the subject is not suitable to participate in this clinical study due to other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Objective Response Rate (ORR) Based on Investigator Assessment Following Treatment in Participants With HER2 alterations Non-Small-Cell Lung Cancer (NSCLC) | Up to 24 months (data cut-off)
  Percentage of Participants who have a complete response (CR) or partial response (PR) as assessed by investigator according to RECIST 1.1

SECONDARY OUTCOMES:
Disease control rate (DCR) Following Treatment in Participants With HER2 alterations Non-Small-Cell Lung Cancer (NSCLC) | Up to 24 months (data cut-off)
  Defined as the proportion of participants who have a complete response (CR), partial response (PR) or standard disease (SD) as assessed by investigator according to RECIST 1.1
Progression-free survival (PFS) Following Treatment in Participants With HER2 alterations Non-Small-Cell Lung Cancer (NSCLC) | Up to 24 months (data cut-off)
  Defined as time from randomization until progression per RECIST 1.1 as assessed by investigator, or death due to any cause.
Duration of Response (DoR) Following Treatment in Participants With HER2 alterations Non-Small-Cell Lung Cancer (NSCLC) | Up to 24 months (data cut-off)
  Defined as the time from the date of first documented response until date of documented progression as assessed by investigator assessment according to RECIST 1.1.
Overall Survival (OS) Following Treatment in Participants With HER2 alterations Non-Small-Cell Lung Cancer (NSCLC) | Up to 24 months (data cut-off)
  Defined as time from randomization until the date of death due to any cause.